## Analytic Plan

Feasibility and Acceptability of a Values-Affirmation Intervention Targeting Medication Adherence in Older Adults with Heart Failure

NCT05310877

1/31/2022

Analysis of the Primary Endpoints: We will examine descriptive statistics (i.e., means, standard deviations, frequencies, percentages) to assess the primary endpoints. Means and standard deviations will be used to describe continuous variables. Frequencies and percentages will be used to describe categorical data. Framework matrix analysis will be used to examine feedback from a qualitative exit interview to provide information on acceptability of study and intervention procedures. Because this study is primarily designed to test feasibility and acceptability of procedures, the study will not be powered to detect statistical differences in self-reported or objectively monitored medication adherence from baseline to end-of-treatment. No inferential statistics are planned.

<u>Baseline Descriptive Statistics</u>: Descriptive statistics will be calculated (i.e., means, standard deviations, frequencies, percentages) to characterize baseline characteristics and demographics of study participants. No inferential statistics are planned in this single-group trial.

<u>Exploratory Analyses</u>: We will examine descriptive statistics (i.e., means, standard deviations) on self-report medication adherence data to determine whether changes are in the expected direction.